CLINICAL TRIAL: NCT05548465
Title: The Safety and Efficacy of Long-term-opioid-free Anesthesia in Anterior Cervical Surgery: a Prospective Randomized Controlled Trial
Brief Title: Long-term-opioid-free Anesthesia in Anterior Cervical Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WCH20220916
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Long-term-opioid-free Anesthesia
MeSH Terms: interventions — Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-term-opioid-free anesthesia group. (Experimental)
  Interventions: Drug: Remifentanil Hydrochloride
- Long-term-opioid anesthesia group. (Active Comparator)
  Interventions: Drug: Sufentanil Citrate

INTERVENTIONS:
Drug: Remifentanil Hydrochloride — Subjects will receive remifentanil anesthesia for operative analgesia.
  Arms: Long-term-opioid-free anesthesia group.
Drug: Sufentanil Citrate — Subjects will receive sufentanil and remifentanil anesthesia for operative analgesia.
  Arms: Long-term-opioid anesthesia group.

SUMMARY:
We design this randomized controlled trial to explore the safety and efficacy of the long-term-opioid-free anesthesia in anterior cervical surgery, to reduce the dosage of perioperative long-acting opioids and promoting patients'rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing anterior cervical surgery., sign the "informed consent form"
* Age above 18 years old
* ASA Ⅰ-Ⅲ.

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with history of drug abuse, including but not limited to opioids, amphetamines, ketamine, etc
* Allergic to the materials or drugs used in this study.
* Patients with current/previous gastrointestinal bleeding and gastric ulcers;
* Have history of nervous system diseases such as peripheral neuropathy, or psychiatric mental illness.
* Other conditions that the investigators consider unsuitable for participation in the study, such as deaf, Parkinson's disease, and difficult to communication etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative numerical rating scales (NRS) at rest. | Up to 48 hours after operation.
  Resting NRS pain scores at 30 min, 2 h, 6 h, 24 h, 48 h after surgery.

SECONDARY OUTCOMES:
Incidence of post operative nausea and vomiting (PONV). | Up to 30 days after operation.
  The proportion of subjects who experienced PONV.
Postoperative NRS on movement. | Up to 48 hours after operation.
  Postoperative NRS pain score on movement, up to 48hr.
Postoperative complications. | Up to 30 days after operation.
  Incidence of postoperative adverse reactions and complications.
Incidence of intraoperative adverse events. | Intraoperative .
Postoperative recovery of cervical spine function | Up to 48 hours after operation.
  Japanese Orthopaedic Association Scores.(JOA scores).
Analgesic medication use before discharge。 | Up to 48 hours after operation.
Length of stay (LOS) in hospital | Up to 30 days after operation.
  Time frame from the day of hospital admission to discharge from the hospital (unit: days).
Postoperative LOS | Up to 30 days after operation.
  Time frame from the day of operation to discharge from the hospital (unit: days).
Total in-hospital cost. | Up to 30 days after operation.
  Total hospitalization expenses after the destruction of costly consumables in orthopedic operation.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D, Principal Investigator — West China Hospital
Locations (1):
- Department of Anesthesiology, West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No